CLINICAL TRIAL: NCT04138004
Title: Comparison of Colon Preparation With 2-Litre Polyethylene Glycol (PEG) Split-dose in Combination With Lubiprostone Versus 4-Litre Polyethylene Glycol (PEG) Split-dose: a Randomized Controlled Trial
Brief Title: Colon Preparation With 2L PEG in Combination With Lubiprostone vs 4L PEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 106/2562
Record Dates: First submitted 2019-10-14; First posted 2019-10-24 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Indication for Modification of Patient Status (Diagnosis)
Keywords: colonoscopy; polyethylene glycols; lubiprostone
MeSH Terms: conditions — Disease | interventions — Polyethylene Glycols; Lubiprostone

STUDY DESIGN:
Intervention Model Description: The research coordinator used a computer to generate a randomization table with blocks of 8. Allocation concealment was maintained through the use of consecutively numbered sealed envelopes. The allocation ratio was 1:1 in 2-L PEG with LB (Group A) or 4-L PEG (Group B). An endoscopy nurse assigned patients to their group and instructed them on the proper use of their assigned bowel preparation method as well as dietary advice.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Gastroenterologists and investigators were blinded to the allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-L PEG with LB (Experimental): PEG used in the present study was Niflec® (Meiji, Japan), which composed of macrogol 4,000 plus electrolytes (sodium sulfate, sodium hydrogen carbonate, sodium chloride, and potassium chloride) and is taken by diluting one sachet into 2-L of plain water. The patients were instructed to take 250 mL every 15 min untill the entire solution was consumed.
  In this group (2-L PEG), half dose preparation started in the evening of the pre-procedure day at about 8.00 to 9.00 pm and the remaining dose was given in the morning at about 5.00 to 6.00 am on the procedure day. And these patients, one 24 mcg tablet of LB was given 2 hours before PEG ingestion (at 6.00 pm of the pre-procedure day).
  Interventions: Drug: polyethylene glycol in combination with lubiprostone
- 4-L PEG (Active Comparator): In this group (4-L PEG), half dose preparation started in the evening of the pre-procedure day at about 8.00 to 10.00 pm and the remaining dose was given in the morning at about 5.00 to 7.00 am on the procedure day.
  Interventions: Drug: polyethylene glycol alone

INTERVENTIONS:
Drug: polyethylene glycol in combination with lubiprostone — 2-litre polyethylene glycol split-dose in combination with one 24 mcg tablet of lubiprostone
  Other Names: NIFLEC in combination with Amitiza
  Arms: 2-L PEG with LB
Drug: polyethylene glycol alone — 4-litre polyethylene glycol split-dose
  Other Names: NIFLEC alone
  Arms: 4-L PEG

SUMMARY:
Colonoscopy is the current standard method for examination of the colon. Bowel cleansing prior to colonoscopy is the essential prerequisite to ensure complete mucosal visualization and lesion identification.(1,2) Suboptimal preparations are associated with missed diagnoses, longer procedure times and increased costs related to the repeat procedures and shortened intervals between procedures.(3-5) Inadequate preparations have been noted in around 25 % cases in the US.(4,6) This has been attributed primarily to poor patient tolerance to the standard colon preparations.

Osmotically balanced polyethylene glycol (PEG) electrolyte bowel lavage solutions were introduced in 1980.(7) These PEG based solutions are the most commonly used bowel preparations today.(7) They have high efficacy, are safe and are associated with minimal fluid and electrolyte imbalance. However the major drawback of these preparations is the taste and the large volumes required with associated nausea, cramping and vomiting.(8) This often results in poor compliance and tolerance with resultant poor preparation and improper visualization. A pooled analysis of 15 trials found that at least 29 % of patients were unable to complete their PEG solution.(9) Lubiprostone (LB) is a locally acting selective Type 2 chloride channel activator which causes intestinal fluid secretion. This results in increased softened stool and increased intestinal transit without the loss of either net intravascular fluid or electrolytes.(10) Peak plasma levels occur approximately 1.14 h after oral administration of a single 24 microgram dose, and the half-life of lubiprostone (t½) has been estimated at approximately 3 h.(11,12) LB is currently approved for the treatment of chronic idiopathic constipation and is generally well tolerated with an excellent side effect profile. Even long term usage has not shown clinically significant changes in electrolyte levels.(10,13) Our hypothesis was that administration of LB in addition to low volume (2-L) split-dose PEG would improve the adequacy of the bowel preparation as comparable as standard 4-L split-dose PEG regimens. Additionally, it could improve patient tolerability and decreased side effects related to the large volume of PEG regimens. Accordingly, we conducted this prospective, single-blind, randomized controlled trial.

DETAILED DESCRIPTION:
Study design:

This was a single center prospective, single-blind, randomized controlled trial to compare the quality of bowel preparation using 2-L PEG with LB vs. 4-L PEG conducted from September 2019 to June 2020 at Department of Medicine, Rajavithi Hospital, a tertiary referral center in Bangkok, Thailand. It was performed in accordance with the clinical principles laid down in the Declaration of Helsinki and informed consent was obtained from all the participants before their enrollment. The study protocol was reviewed and approved by the ethics committee of Rajavithi Hospital. Recruitment, enrollment, randomization, withdrawal, and completion were done according to the consort guidelines.

Bowel preparation method:

PEG used in the present study was Niflec® (Meiji, Japan), which composed of macrogol 4,000 plus electrolytes (sodium sulfate, sodium hydrogen carbonate, sodium chloride, and potassium chloride) and is taken by diluting one sachet into 2-L of plain water. The participants were instructed to take 250 mL every 15 min untill the entire solution was consumed. In cases of 4-L split-dosage, half dose preparation started in the evening of the pre-procedure day at about 8.00 to 10.00 pm and the remaining dose was given in the morning at about 5.00 to 7.00 am on the procedure day. In cases of 2-L split-dosage, half dose preparation started in the evening of the pre-procedure day at about 8.00 to 9.00 pm and the remaining dose was given in the morning at about 5.00 to 6.00 am on the procedure day. And these patients, one 24 mcg tablet of LB was given 2 hours before PEG ingestion (at 6.00 pm of the pre-procedure day).

Dietary advice was given to all patients. Consumption of fruit, legumes, or vegetable was forbidden 2 days before the procedure. On the day before colonoscopy patients had a light breakfast and lunch, but a liquid dinner (clear soup). Solid food was not allowed at the start of the bowel preparation phase. All patients were instructed to fast from midnight before procedure day, but some anti-hypertensive drugs and minimal plain water were permitted.

Randomization:

All participants attended an informational session before colonoscopy where the participants were counseled about the nature of the study and written informed consent was obtained. The research coordinator used a computer to generate a randomization table with blocks of 8. Allocation concealment was maintained through the use of consecutively numbered sealed envelopes. The allocation ratio was 1:1 in 2-L PEG with LB (Group A) or 4-L PEG (Group B).

An endoscopy nurse assigned the participants to their group and instructed the participants on the proper use of their assigned bowel preparation method as well as dietary advice. Gastroenterologists and investigators were blinded to the allocation groups. The participants were given a questionnaire measured the tolerability and side effects of the bowel preparation regimen, to be completed once their bowel preparation was finished and before coming to the hospital for the colonoscopy.

Colonoscopy:

All colonoscopies were performed by 3 experienced gastroenterologists (minimum experience of 1000 procedures; Apichet Sirinawasatien, Kanokpoj Chanpiwat, and Tanyaporn Chantarojanasiri) at the Rajavithi Hospital. A standard protocol for insertion, withdrawal, and observation was followed. All colonoscopies were performed using video colonoscopes (CF 180, Olympus, Japan) under moderate sedation.

The colon segment including the rectum and extending up to the splenic flexure was termed as left colon; the segment between splenic flexure and hepatic flexure was termed transverse colon; while colon segment proximal to hepatic flexure, including the cecum was termed right colon for the purpose of this study. A complete colonoscopy was defined as reaching the cecum determined by the visualization and documentation of the ileocecal valve and appendiceal orifice. Failed colonoscopy was defined as endoscope could not reach ileocecal valve and cecum. Overall procedure times was the times between the endoscope enter and withdraw from the anus.

During the insertion of the scope, two representative pictures were taken from each of these three segments to document the colon preparation. An early colonoscopy was defined as a procedure initiated during 8-11 am while those started after 11 am were considered the late procedure.

Colon cleansing scale:

The investigators used Boston bowel preparation scale (BBPS) score to evaluate the adequacy of the preparation. Each colonic segment was graded from 0 (solid stools) to 3 (no residual staining). The aggregate score was obtained by adding the score for all 3 segments, thus resulting in a score between 0 and 9. A score ≤4 was considered a poor colon preparation, resulting in a recommendation for a repeat procedure. A score of 8-9 was considered excellent preparation while a score of 5-7 was considered adequate preparation.

The colon preparation was graded by analyzing photo documentation obtained during a colonoscopy by three gastroenterologists (AS, KC, and TC) after the procedure finished. The mean BBPS score of each patient was calculated and recorded the result on a separate standardized form.

Sample size calculation and statistical analysis:

Descriptive statistics were used for baseline characteristics. The Boston bowel preparation scale produces data that are approximately normally distributed. Two-group ANOVA was used to assess for the presence of group differences in the preparation scores while accounting for procedure time (early versus late). The proportion of adequate bowel preparation in each group was compared with a chi-square statistic. The secondary endpoints of tolerability and side effects were assessed using the Mann-Whitney U test.

The sample size was calculated using two independent means formula (two-tailed test) based on data from a previous study in 2008,(16) in which the patient mean overall symptom questionnaire ratings of the PEG plus LB group was 3.7±1 compared to 3.2±1.1 in the controlled group (p = 0.003). The minimum required number of participants was calculated at 70 in each group in order to detect a signiﬁcant association with 80% power (β =0.20) and a 5% probability of type I error (2-sided) (α =0.05).

ELIGIBILITY:
Inclusion Criteria:

* All patients between the age of 18 and 75 years with an appropriate indication for elective colonoscopy were considered eligible.

Exclusion Criteria:

* We excluded patients who (i) suspected gastroparesis, gastric outlet or bowel obstruction; (ii) had a previous history of any gastrointestinal surgery apart from an appendectomy and cholecystectomy; (iii) had severe cardiac or pulmonary disease (American Society of Anesthesiologists physical status class 3 or 4), severe renal failure (creatinine clearance <30 mL/min), decompensated liver cirrhosis or severe systemic illness; (iv) had a compromised swallowing reflex or impaired mental status; (v) were in a state of pregnancy or lactating; (vi) were hypersensitive or allergic to PEG or LB; or (vii) had a history of previous failure of adequate bowel preparation for colonoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
the degree of colon cleansing | up to 7 months
  We used Boston bowel preparation scale (BBPS) score to evaluate the adequacy of the preparation. Each colonic segment was graded from 0 (solid stools) to 3 (no residual staining). The aggregate score was obtained by adding the score for all 3 segments, thus resulting in a score between 0 and 9. A score ≤4 was considered a poor colon preparation, resulting in a recommendation for a repeat procedure. A score of 8-9 was considered excellent preparation while a score of 5-7 was considered adequate preparation.
  The colon preparation was graded by analyzing photo documentation obtained during a colonoscopy by three gastroenterologists (AS, KJ, and TC) after the procedure finished. The mean BBPS score of each patient was calculated and recorded the result on a separate standardized form.

SECONDARY OUTCOMES:
patient's tolerability | up to 7 months
  The patient's tolerability on taking the bowel preparation was evaluated with a 10-cm visual analog scale which 10 means excellent and 0 means very poor.
adverse events related to bowel preparation | up to 7 months
  Any adverse events related to bowel preparation (nausea, vomiting, bloating, abdominal pain, dizziness, etc.) were recorded by the endoscopy nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Apichet Sirinawasatien, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jemal A, Center MM, DeSantis C, Ward EM. Global patterns of cancer incidence and mortality rates and trends. Cancer Epidemiol Biomarkers Prev. 2010 Aug;19(8):1893-907. doi: 10.1158/1055-9965.EPI-10-0437. Epub 2010 Jul 20. PMID 20647400
- [Result] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Result] Bae SE, Kim KJ, Eum JB, Yang DH, Ye BD, Byeon JS, Myung SJ, Yang SK, Kim JH. A Comparison of 2 L of Polyethylene Glycol and 45 mL of Sodium Phosphate versus 4 L of Polyethylene Glycol for Bowel Cleansing: A Prospective Randomized Trial. Gut Liver. 2013 Jul;7(4):423-9. doi: 10.5009/gnl.2013.7.4.423. Epub 2013 Jun 11. PMID 23898382
- [Result] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Result] Seeff LC, Nadel MR, Klabunde CN, Thompson T, Shapiro JA, Vernon SW, Coates RJ. Patterns and predictors of colorectal cancer test use in the adult U.S. population. Cancer. 2004 May 15;100(10):2093-103. doi: 10.1002/cncr.20276. PMID 15139050
- [Result] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Result] Davis GR, Santa Ana CA, Morawski SG, Fordtran JS. Development of a lavage solution associated with minimal water and electrolyte absorption or secretion. Gastroenterology. 1980 May;78(5 Pt 1):991-5. PMID 7380204
- [Result] Adamcewicz M, Bearelly D, Porat G, Friedenberg FK. Mechanism of action and toxicities of purgatives used for colonoscopy preparation. Expert Opin Drug Metab Toxicol. 2011 Jan;7(1):89-101. doi: 10.1517/17425255.2011.542411. PMID 21162694
- [Result] Tan JJ, Tjandra JJ. Which is the optimal bowel preparation for colonoscopy - a meta-analysis. Colorectal Dis. 2006 May;8(4):247-58. doi: 10.1111/j.1463-1318.2006.00970.x. PMID 16630226
- [Result] Lacy BE, Levy LC. Lubiprostone: a chloride channel activator. J Clin Gastroenterol. 2007 Apr;41(4):345-51. doi: 10.1097/01.mcg.0000225665.68920.df. PMID 17413599
- [Result] Lacy BE, Levy LC. Lubiprostone: a novel treatment for chronic constipation. Clin Interv Aging. 2008;3(2):357-64. doi: 10.2147/cia.s2938. PMID 18686757
- [Result] Owen RT. Lubiprostone--a novel treatment for irritable bowel syndrome with constipation. Drugs Today (Barc). 2008 Sep;44(9):645-52. doi: 10.1358/dot.2008.44.9.1269852. PMID 19137119
- [Result] Grigg E, Schubert MC, Hall J, Rahhal F, Raina D, Sridhar S, Chamberlain SM. Lubiprostone used with polyethylene glycol in diabetic patients enhances colonoscopy preparation quality. World J Gastrointest Endosc. 2010 Jul 16;2(7):263-7. doi: 10.4253/wjge.v2.i7.263. PMID 21160617
- [Result] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Result] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Result] Stengel JZ, Jones DP. Single-dose lubiprostone along with split-dose PEG solution without dietary restrictions for bowel cleansing prior to colonoscopy: a randomized, double-blind, placebo-controlled trial. Am J Gastroenterol. 2008 Sep;103(9):2224-30. doi: 10.1111/j.1572-0241.2008.02053.x. Epub 2008 Aug 5. PMID 18684185